CLINICAL TRIAL: NCT04386811
Title: Vitamin D as a Therapeutic Adjunct in the Stimulant Treatment of ADHD: a Proof-of-concept Tele-health Study of Stimulant-induced Improvement in Neurocognitive Functioning.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Following Yale University resuming in-person research activities, the investigators no longer had dedicated funding for the study and were unable to secure additional funding to meet the research goals.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2000028035
Record Dates: First submitted 2020-05-07; First posted 2020-05-13 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Calcitriol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Calcitriol (Experimental)
  Interventions: Drug: Calcitriol
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Calcitriol — A total of 24 otherwise medically healthy individuals with ADHD will be studied as outpatients. All subjects will undergo neurocognitive assessments of attention/vigilance, spatial working memory, and reversal learning both before and after subjects' daily dosing with their currently prescribed stimulant medication on both calcitriol and placebo pretreatment days using a randomized, double-blind, placebo controlled, within-subject, two-day study design.
  Arms: Calcitriol
Other: Placebo — A total of 24 otherwise medically healthy individuals with ADHD will be studied as outpatients. All subjects will undergo neurocognitive assessments of attention/vigilance, spatial working memory, and reversal learning both before and after subjects' daily dosing with their currently prescribed stimulant medication on both calcitriol and placebo pretreatment days using a randomized, double-blind, placebo controlled, within-subject, two-day study design.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess vitamin D as a therapeutic adjunct in the stimulant treatment of ADHD.

DETAILED DESCRIPTION:
The specific aim of this study is to determine whether acute calcitriol (vitaminD) administration (compared to placebo) enhances the neurocognitive effects of of current stimulant medications as measured by tasks of vigilance/attention, spatial working memory, and reversal learning in individuals with (attention deficit hyperactivity disorder (ADHD) using a randomized, double-blind, placebo controlled, within-subject, two-day study design.

Primary Hypothesis: It is hypothesized that calcitriol (versus placebo) administration will enhance positive neurocognitive effects of current stimulant medications in individuals with ADHD.

Secondary (Exploratory) Hypothesis: It is hypothesized that calcitriol (versus placebo) administration alone will also enhance neurocognitive performance on tasks of attention/vigilance and/or spatial working memory.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years
* Voluntary, written, informed consent
* Physically healthy by medical and psychiatric history
* DSM-5 diagnosis of ADHD
* Point of Care Test results for Vitamin D equal or higher than 20 ng/ml
* English speaking

Exclusion Criteria:

* Medical contraindication to calcitriol administration (e.g., history of hypersensitivity to calcitriol or any component of the formulation, hypercalcemia or vitamin D toxicity)
* History of substance dependence (e.g., alcohol, opiates, sedative hypnotics), except for nicotine
* A primary major DSM-V psychiatric disorder (e.g., schizophrenia, bipolar disorder, major depression, etc.) as determined by the Structured Clinical Interview for DSM-V (SCID), except ADHD
* A history of significant medical (e.g., cardiovascular, diabetic/metabolic) or neurological (e.g., cerebrovascular accidents, seizure, traumatic brain injury) illness
* Current use of psychotropic and/or potentially psychoactive prescription medications, except prescribed stimulants
* Use of any prescription medications and/or over-the-counter medications, vitamins (including vitamin D) and/or herbal supplements which could have a negative clinical interaction with calcitriol or which could confound scientific results of the study, within 2 weeks prior to each test day (e.g., thiazide diuretics, Mg based antiacids, digoxin, etc,).
* Levels of 25(OH)D3 below 20 ng/ml .
* History of kidney stones within the past 5 years
* History of renal failure
* History of parathyroid disorder (hyper or hypoparathyroidism)
* History of osteoporosis or any pathologic fractures
* Vitamin D supplementation in any form in the past 3 months
* Known hypersensitivity to calcitriol
* Malabsorption syndromes (i.e. Celiac sprue)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
Enhanced positive neurocognitive effects on the CPT-IP | Up to 5 hours
  On the Continuous Performance Task (CPT-IP) subjects are shown a random sequence of different numbers and are instructed to press a button as quickly and accurately as possible upon detection of two identical pairs of numbers, and to withhold their response to any other sequence of letters. Outcomes will be measured by d prime.
Enhanced positive neurocognitive effects on the Spatial working memory task | Up to 5 hours
  The spatial working memory task is a measure of working memory. As part of the task, stimuli will be projected onto the computer screen and target stimuli can be spatial locations, different visual stimuli, sound or text. Outcomes will be measured by percent correct.
Enhanced positive neurocognitive effects on the PRLT | Up to 5 hours
  The Probabilistic Reversal Learning Task (PRLT) measures subjects' perseverative responding in the context of changing reward contingencies / cues. Outcomes will be measured by numbers of reversal achieved, total points, and error types.

SECONDARY OUTCOMES:
Enhanced positive neurocognitive effects on the CPT-IP- hits | Up to 5 hours
  Enhanced positive neurocognitive effects on the CPT-IP will be measured by counts of hits, false alarms, and random errors.
Enhanced positive neurocognitive effects on the CPT-IP- false alarms | Up to 5 hours
  Enhanced positive neurocognitive effects on the CPT-IP will be measured by counts of hits, false alarms, and random errors.
Enhanced positive neurocognitive effects on the CPT-IP- random errors | Up to 5 hours
  Enhanced positive neurocognitive effects on the CPT-IP will be measured by counts of hits, false alarms, and random errors.Enhanced positive neurocognitive effects on the CPT-IP will be measured by counts of hits, false alarms, and random errors.Enhanced positive neurocognitive effects on the CPT-IP will be measured by counts of hits, false alarms, and random errors.
Spatial working memory task- reaction time | Up to 5 hours
  Enhanced positive neurocognitive effects be measured by reaction time on the spatial working memory task.
Enhanced positive neurocognitive effects on the PRLT - win-switch / lose-stay rate | Up to 5 hours
  Enhanced positive neurocognitive effects on the PRLT will be measured by win-switch / lose-stay rate.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Potenza, MD, Principal Investigator — Yale University
Locations (1):
- CMHC, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided